CLINICAL TRIAL: NCT00548548
Title: A Double-blind, Randomised, Multicenter, Phase III Study of Bevacizumab in Combination With Capecitabine and Cisplatin Versus Placebo in Combination With Capecitabine and Cisplatin, as First-line Therapy in Patients With Advanced Gastric Cancer
Brief Title: A Study of Bevacizumab in Combination With Capecitabine and Cisplatin as First-line Therapy in Patients With Advanced Gastric Cancer
Acronym: AVAGAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry); Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF4200g; BO20904 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Adenocarcinoma
Keywords: Avastin; Metastatic Adenocarcinoma; AVAGAST
MeSH Terms: conditions — Adenocarcinoma | interventions — Bevacizumab; Capecitabine; Cisplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab (Experimental): Participants received intravenous (IV) bevacizumab 7.5 mg/kg every 3 weeks, oral capecitabine 1,000 mg/m˄2 twice daily for 14 days every 3 weeks, or 5-fluorouracil (5-FU) at a dose of 800 mg/m˄2/day as a continuous IV infusion over the first 5 days of every 3 week cycle, and cisplatin 80 mg/m˄2 as an IV infusion every 3 weeks for a maximum of 6 cycles. Bevacizumab and capecitabine/5-FU were administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Cisplatin; Drug: 5-fluorouracil
- Placebo (Placebo Comparator): Participants received intravenous (IV) placebo infusion every 3 weeks, oral capecitabine 1,000 mg/m˄2 twice daily for 14 days every 3 weeks, or 5-fluorouracil (5-FU) at a dose of 800 mg/m˄2/day as a continuous IV infusion over the first 5 days of every 3 week cycle, and cisplatin 80 mg/m˄2 as an IV infusion every 3 weeks for a maximum of 6 cycles. The placebo and capecitabine/5-FU were administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Placebo; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Bevacizumab — Intravenous bevacizumab 7.5 mg/kg once every 3 weeks, given until disease progression or unmanageable toxicity.
  Arms: Bevacizumab
Drug: Capecitabine — Oral capecitabine 1,000 mg/m˄2 twice daily for 14 days every 3 weeks, given until disease progression or unmanageable toxicity.
Drug: Cisplatin — Cisplatin 80 mg/m˄2 as a 2 hr intravenous infusion with hyper-hydration and pre-medication (steroids and anti-emetics), given every 3 weeks for a maximum of 6 cycles or until disease progression or unmanageable toxicity.
Drug: Placebo — Intravenous placebo every 3 weeks, given until disease progression or unmanageable toxicity.
  Arms: Placebo
Drug: 5-fluorouracil — For participants with difficulty swallowing, malabsorption, or other conditions that could affect intake of oral capecitabine medication, 5-fluorouracil was administered instead, at a dose of 800 mg/m˄2/day as a continuous intravenous infusion over 5 days (days 1 to 5 of each cycle), every 3 weeks.

SUMMARY:
This study will compare treatment with bevacizumab in combination with capecitabine and cisplatin versus placebo in combination with capecitabine and cisplatin, as first-line therapy in patients with locally advanced or metastatic gastric cancer who had not received prior chemotherapy for advanced or metastatic disease.

DETAILED DESCRIPTION:
This is a 2 arm, randomized, double-blind, multicenter phase III study. Patients will be randomized (1:1) to capecitabine/cisplatin plus bevacizumab or capecitabine/cisplatin plus placebo. This is an event-driven trial with the primary analysis planned after approximately 517 deaths had been observed. After the primary analysis, the study will remain open and patients can continue with study treatment until progressive disease or earlier at the investigator's discretion. After discontinuation of the last patient, the study will end globally.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study specific procedures.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Life expectancy of at least 3 months.
* Able to comply with the protocol.
* Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable, locally advanced, or metastatic disease, not amenable to curative therapy.
* Measurable disease or non-measurable but evaluable disease, according to the Response Evaluation Criteria in Solid Tumours (RECIST).
* Patient not receiving anticoagulant medication must have an International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 x Upper Limit of Normal (ULN) within 7 days prior to randomisation.

Exclusion Criteria:

* Previous chemotherapy for locally advanced or metastatic gastric cancer. Patients may have received prior neoadjuvant or adjuvant chemotherapy as long as it was completed at least 6 months prior to randomisation.
* Previous platinum or anti-angiogenic therapy (ie, anti-vascular endothelial growth factor [VEGF] or VEGF receptor tyrosine kinase inhibitor, etc.).
* Patients with locally advanced disease who are candidates for curative therapy (including operation and/or chemotherapy and/or radiotherapy).
* Radiotherapy within 28 days of randomisation.
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomisation, or anticipation of the need for major surgery during the course of the study treatment (planned elective surgery).
* Minor surgical procedures within 2 days prior to randomisation.
* Evidence of central nervous system (CNS) metastasis at baseline.
* History or evidence upon physical/neurological examination of CNS disease unrelated to cancer unless adequately treated with standard medical therapy, eg, uncontrolled seizures.
* History of another malignancy which could affect compliance with the protocol or interpretation of results.
* Inadequate bone marrow function.
* Inadequate liver function.
* Inadequate renal function.
* Uncontrolled hypertension or clinically significant (ie, active) cardiovascular disease.
* Active infection requiring intravenous antibiotics at randomisation.
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Serious or non-healing wound, peptic ulcer, or (incompletely healed) bone fracture.
* Active gastrointestinal bleeding.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of randomisation.
* Neuropathy (eg, impairment of hearing and balance) ≥ grade II according to Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
* Chronic daily treatment with aspirin or clopidogrel.
* Chronic daily treatment with oral corticosteroids; inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed.
* Known hypersensitivity to any of the study drugs or excipients or to Chinese hamster ovary cell products or to other recombinant human or humanised antibodies.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Evidence of any other disease, metabolic or psychological dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or that may affect patient compliance with the study, or place the patient at high risk from treatment complications.
* Known acute or chronic-active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Pregnant or lactating females.
* Women of childbearing potential not using effective nonhormonal (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly, or surgically sterile) means of contraception.
* Sexually active men unwilling to practice contraception during the study.
* Current or recent (within the 28 days prior to randomisation) treatment with another investigational drug or participation in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hedrick, MD, Study Director — Genentech, Inc.
Locations (13):
- United States (13):
  - Tower Cancer Research Fnd, Beverly Hills, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Kenmar Research Institute LLC, Los Angeles, California
  - USC/Norris Cancer Center, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - H. Lee Moffitt Cancer, Tampa, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Methodist Cancer Center Onc, Omaha, Nebraska
  - Memorial Sloan Kettering, New York, New York
  - Duke Univ Medical Center, Durham, North Carolina
  - South Carolina Oncology Assoc, Columbia, South Carolina
  - The Sarah Cannon Research Inst, Nashville, Tennessee

REFERENCES:
- [Derived] Han K, Jin J, Maia M, Lowe J, Sersch MA, Allison DE. Lower exposure and faster clearance of bevacizumab in gastric cancer and the impact of patient variables: analysis of individual data from AVAGAST phase III trial. AAPS J. 2014 Sep;16(5):1056-63. doi: 10.1208/s12248-014-9631-6. Epub 2014 Jun 19. PMID 24942210
- [Derived] Ohtsu A, Shah MA, Van Cutsem E, Rha SY, Sawaki A, Park SR, Lim HY, Yamada Y, Wu J, Langer B, Starnawski M, Kang YK. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a randomized, double-blind, placebo-controlled phase III study. J Clin Oncol. 2011 Oct 20;29(30):3968-76. doi: 10.1200/JCO.2011.36.2236. Epub 2011 Aug 15. PMID 21844504

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab | Placebo
Started | 387 | 387
Treated | 383 | 384
Safety Population | 386 (Four patients randomized to placebo received single doses of bevacizumab in error.) | 381
Completed | 25 (Completed treatment discontinuation form was not completed; patient was counted alive on treatment.) | 21
Not Completed | 362 | 366
Not completed — Death | 345 | 348
Not completed — Lost to Follow-up | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Placebo | Total
Number analyzed (Participants) | 387 | 387 | 774
Age, Customized [Number; unit: participants]
  <40 | 36 | 29 | 65
  40-65 | 241 | 249 | 490
  ≥65 | 110 | 109 | 219
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 129 | 259
  Male | 257 | 258 | 515

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary efficacy endpoint for this study was overall survival (time to death), defined as the time between randomization and the date of death irrespective of the cause of death. Patients for whom no death was captured on the clinical database were censored at the most recent date they were known to be alive. Median survival was estimated by the Kaplan-Meier method.
Time Frame: From randomization until death, up to 26 months
Population: The Intent-to-Treat population, including all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 387 | 387
months | 12.1 [11.1 to 13.8] | 10.1 [9.0 to 11.3]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time between randomization and the date of first documented disease progression or death, whichever occurs first. Patients who neither progressed nor died at the time of study completion or who were lost to follow-up were censored at the date of the last tumor assessment or last follow up for progression of disease. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From randomization until disease progression or death, up to 26 months.
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 387 | 387
months | 6.7 [5.9 to 7.1] | 5.3 [4.4 to 5.6]

3. Secondary Outcome: Progression-free Survival During First-line Therapy
Description: Progression-free survival (PFS) during first-line therapy is defined as the time between randomization and the date of first documented disease progression or death, whichever occurs first and only if it occurs no later than 28 days after last confirmed intake of any study medication and only if it occurs before the start of non-study antineoplastic treatment. Participants who did not progress or die in this interval or were lost to follow-up were censored at the date of the last tumor assessment within this time window. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From randomization until 28-days after the last study treatment was administered, up to 26 months.
Population: Intent-to treat.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 387 | 387
months | 6.9 [6.2 to 7.3] | 5.4 [4.7 to 5.6]

4. Secondary Outcome: Time to Disease Progression
Description: Time to progression is defined as the time from randomization to the first occurrence of progressive disease (PD). PD was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions, or appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Patients with no PD at study completion (including those who died before PD) were censored at the date of the last tumor assessment. Median time to PD was estimated using the Kaplan-Meier method.
Time Frame: From randomization until disease progression; assessed every 6 weeks for the first year and every 12 weeks thereafter, up to 26 months.
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 387 | 387
months | 7.0 [6.5 to 7.6] | 5.6 [5.1 to 5.8]

5. Secondary Outcome: Participants With a Best Overall Response of Complete or Partial Response
Description: Best overall response during first-line therapy is defined as the occurrence of either a confirmed complete (CR) or a partial (PR) best overall response, as determined by the RECIST criteria. CR is defined as the disappearance of all target and non-target lesions and PR is defined as at least a 30% decrease in the sum of the longest diameter of target lesions and no new or progression of non-target lesions, or the disappearance of all target lesions and persistence of one or more non-target lesion(s).
Time Frame: From randomization until the end of study, up to 26 months.
Population: Measurable Disease Population, including all randomized participants with measurable disease (per RECIST) for gastric cancer at baseline. Patients were analyzed according to the treatment groups to which they were randomized.
Measure: Number; unit: participants
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 311 | 297
participants
  Responders | 143 | 111
  Non-responders | 168 | 186

6. Secondary Outcome: Duration of Response
Description: Duration of response during first line therapy is defined as the time from when response (CR or PR) was first documented to first documented disease progression or death (whichever occurs first) during first line therapy. This was only be calculated for participants who achieved a best overall response of CR or PR. Participants who did not progress or die after they had a confirmed response were censored at the date of their last tumor measurement or last follow up for progression of disease during first line therapy. Median duration of response was estimated using the Kaplan-Meier method.
Time Frame: From randomization to the end of study, up to 26 months
Population: Participants with measurable disease at baseline who had a best overall response of complete response or partial response, and for whom duration of response data was available.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 142 | 111
months | 7.1 [6.2 to 8.3] | 5.8 [4.6 to 6.9]

7. Secondary Outcome: Participants With Disease Control
Description: Disease control for participants with measurable disease was defined as a complete response (CR), partial response (PR) or stable disease (SD) for 6 weeks or longer, as determined by the RECIST criteria. For participants without measurable disease, disease control was defined as no disease progression for ≥ 6 weeks.
Time Frame: From randomization until the end of study, up to 26 months.
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 387 | 387
participants
  Participants with Disease Control | 300 | 271
  Participants without Disease Control | 87 | 116

8. Secondary Outcome: Participants With Adverse Events
Description: The intensity of Adverse Events (AEs) was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3.0 on a five-point scale from Grade 1 (Mild) to Grade 5 (Death). A serious AE (SAE) was defined as any event that is fatal, life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From randomization until 3 months after last dose (up to 26 months)
Population: Safety population, including all patients randomized and exposed to study medication (defined as any one component of the combination). Patients are assigned to treatment groups based on the treatment they actually received.
Measure: Number; unit: participants
Arm/Group | Bevacizumab | Placebo
Number analyzed (Participants) | 386 | 381
participants
  Any Adverse event | 380 | 377
  Serious AE | 134 | 137
  Grade 3/4/5 AE | 293 | 294
  Grade 5 AE | 18 | 25
  Deaths not due to Progression | 31 | 29

ADVERSE EVENTS:
Time Frame: From time of very first drug intake until 91 day(s) after very last drug intake.
Description: Safety population: All randomized participants who were exposed to study medication (defined as any one component of the combination).
Arm/Group | Bevacizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 134/386 | 137/381
Other Adverse Events (participants affected / at risk) | 378/386 | 373/381
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=386) | Placebo (N=381)
VOMITING (Gastrointestinal disorders) | 11 | 18
DIARRHOEA (Gastrointestinal disorders) | 16 | 8
NAUSEA (Gastrointestinal disorders) | 7 | 12
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 5
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 5 | 4
GASTRIC PERFORATION (Gastrointestinal disorders) | 7 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 2
DYSPHAGIA (Gastrointestinal disorders) | 1 | 3
STOMATITIS (Gastrointestinal disorders) | 3 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 2
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 1 | 1
ILEUS (Gastrointestinal disorders) | 1 | 1
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 | 1
PERITONITIS (Infections and infestations) | 1 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 1 | 0
DUODENAL PERFORATION (Gastrointestinal disorders) | 0 | 1
ENTERITIS (Gastrointestinal disorders) | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 1
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 1 | 0
GASTRIC STENOSIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
ILEAL PERFORATION (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 13 | 13
NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 10
ANAEMIA (Blood and lymphatic system disorders) | 6 | 7
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 3
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 1
MICROANGIOPATHIC HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 | 13
DEHYDRATION (Metabolism and nutrition disorders) | 7 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 7
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 8 | 7
SEPSIS (Infections and infestations) | 4 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 2
INFECTION (Infections and infestations) | 2 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 0 | 2
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 1
APPENDICITIS (Infections and infestations) | 0 | 1
BACILLUS INFECTION (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
LUNG ABSCESS (Infections and infestations) | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 1
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 | 0
TOOTH INFECTION (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0
ASTHENIA (General disorders) | 4 | 6
FATIGUE (General disorders) | 5 | 3
DEATH (General disorders) | 3 | 4
PYREXIA (General disorders) | 4 | 3
CHEST PAIN (General disorders) | 2 | 0
ADVERSE DRUG REACTION (General disorders) | 0 | 1
CATHETER THROMBOSIS (General disorders) | 0 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
HYPERPYREXIA (General disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 8 | 13
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 4
HYPERTENSION (Vascular disorders) | 1 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1
HAEMORRHAGE (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 1 | 0
VASOSPASM (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 4 | 3
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 2 | 0
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
RENAL SALT-WASTING SYNDROME (Renal and urinary disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 2
CONVULSION (Nervous system disorders) | 1 | 1
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 2 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 | 0
AFFERENT LOOP SYNDROME (Injury, poisoning and procedural complications) | 0 | 1
DEVICE MALFUNCTION (Injury, poisoning and procedural complications) | 1 | 0
OESOPHAGEAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1
STENT OCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 4
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 0
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 2 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 2 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR NECROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR PERFORATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 1
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 1
BLOOD SODIUM DECREASED (Investigations) | 0 | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 0
RETINOPATHY (Eye disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 0
DEVICE OCCLUSION (General disorders) | 1 | 0
STENT MALFUNCTION (General disorders) | 1 | 0
THROMBOSIS IN DEVICE (General disorders) | 1 | 0
EMBOLISM (Vascular disorders) | 0 | 1
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 | 1
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 1
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
STOMA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=386) | Placebo (N=381)
NAUSEA (Gastrointestinal disorders) | 264 | 248
VOMITING (Gastrointestinal disorders) | 192 | 188
DIARRHOEA (Gastrointestinal disorders) | 180 | 142
CONSTIPATION (Gastrointestinal disorders) | 141 | 124
STOMATITIS (Gastrointestinal disorders) | 111 | 88
ABDOMINAL PAIN (Gastrointestinal disorders) | 82 | 55
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 39 | 32
DYSPEPSIA (Gastrointestinal disorders) | 23 | 16
GINGIVITIS (Infections and infestations) | 25 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 250 | 221
ANAEMIA (Blood and lymphatic system disorders) | 83 | 111
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 70 | 67
LEUKOPENIA (Blood and lymphatic system disorders) | 21 | 18
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 183 | 124
ALOPECIA (Skin and subcutaneous tissue disorders) | 94 | 87
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 56 | 53
RASH (Skin and subcutaneous tissue disorders) | 39 | 32
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 27 | 13
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 22 | 13
FATIGUE (General disorders) | 157 | 145
ASTHENIA (General disorders) | 77 | 64
PYREXIA (General disorders) | 54 | 51
MUCOSAL INFLAMMATION (General disorders) | 53 | 32
OEDEMA PERIPHERAL (General disorders) | 30 | 37
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 55 | 50
HEADACHE (Nervous system disorders) | 51 | 36
NEUROPATHY PERIPHERAL (Nervous system disorders) | 42 | 41
DYSGEUSIA (Nervous system disorders) | 42 | 39
DIZZINESS (Nervous system disorders) | 38 | 41
DECREASED APPETITE (Metabolism and nutrition disorders) | 204 | 175
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 52 | 56
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 64 | 20
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18 | 25
COUGH (Respiratory, thoracic and mediastinal disorders) | 15 | 22
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 49 | 63
WEIGHT DECREASED (Investigations) | 44 | 43
HYPERTENSION (Vascular disorders) | 84 | 51
BACK PAIN (Musculoskeletal and connective tissue disorders) | 29 | 21
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 21 | 7
PROTEINURIA (Renal and urinary disorders) | 28 | 20
RENAL IMPAIRMENT (Renal and urinary disorders) | 24 | 21
INSOMNIA (Psychiatric disorders) | 43 | 37
NASOPHARYNGITIS (Infections and infestations) | 26 | 15
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 24 | 14
HYPOKALAEMIA (Metabolism and nutrition disorders) | 17 | 18
DEHYDRATION (Metabolism and nutrition disorders) | 19 | 11
MYALGIA (Musculoskeletal and connective tissue disorders) | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.